CLINICAL TRIAL: NCT00421447
Title: Bone Geometry and Muscle Density Changes in Postmenopausal Women and Breast Cancer Patients Prescribed Anastrozole
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Professor, McMaster University
Organization: McMaster University (Other)
Other Study IDs: 06-375
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; pQCT; Anastrozole; bone geometry
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast Cancer patients: A group of women with breast cancer prescribed Anastrozole
  Interventions: Drug: Anastrozole
- Healthy women wit no breast Cancer: A group of healthy women wit no breast cancer prescribed Anastrozole
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — Group of women with breast cancer
  Other Names: Anastrozole medication

SUMMARY:
The primary objective of this study is to determine if trabecular or cortical volumetric bone mineral density (vBMD) change over time in postmenopausal breast cancer patients who are prescribed Anastrozole, as measured by pQCT at the proximal and distal radius and tibia.

DETAILED DESCRIPTION:
In bone, where estrogen is required to maintain density, there is indication of increased turnover in patients prescribed Aromatase Inhibitors. However, there are no studies to date that prospectively quantify the impact of Aromatase inhibitors on bone quality. Furthermore, the actual effects and clinical significance of adjuvant chemotherapy and supportive medications on bone quality in women with breast carcinoma is unknown. The current study proposes to prospectively assess novel skeletal health outcomes, namely trabecular structure (connectivity, hole size) and bone geometry (bone area, cortical thickness) among women with breast cancer being treated with Anastrozole. Not only will the current study provide a better understanding of the changes in bone quality and muscle mass after Anastrozole treatment, it will provide important information about the development of secondary skeletal complications in this population. Therefore, the potential to collect data prospectively from a cohort of individuals with breast cancer being treated with Anastrozole represents an important step to advance knowledge in this area. Also, by examining bone quality and secondary complications in a diverse cohort of patients who vary with respect to radiation therapy, chemotherapy and additional medications, we can begin to identify patterns of musculoskeletal change and predictors of these changes.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Treatment Group

* Postmenopausal breast cancer patients (stage 1 and 2)
* Non-institutionalized
* Prescribed Anastrozole within the preceding 1-2 weeks
* Ambulatory
* Ability to read and comprehend study protocol and informed consent

Group 2: Control Group

* Healthy, age-matched postmenopausal women
* Non-institutionalized
* Ambulatory
* Ability to read and comprehend study protocol and informed consent

Exclusion Criteria:

* Prior Tamoxifen or Raloxifene therapy
* Known congenital metabolic bone disease (e.g., osteogenesis imperfecta)
* Concomitant treatment with corticosteroids
* Patients with a history of endocrine disorders or surgical parathyroidectomy
* Patients with disorders known to affect bone metabolism including diabetes mellitus, systemic lupus erythematosus, Cushing's disease, hyperparathyroidism, chronic liver disease, chronic renal failure, Paget's disease
* Conditions preventing pQCT measurement (e.g., unable to lie flat or still for 15 minutes)
* Geographically inaccessible for follow-up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-menopausal Women
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, M.D., Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster University, Hamilton, Ontario, Canada